CLINICAL TRIAL: NCT01509508
Title: A Cluster Randomised Trial Comparing the Impact of Immediate Versus South African Recommendations Guided ART Initiation on HIV Incidence. The ARNS 12249 TasP (Treatment as Prevention) Trial in Hlabisa Sub-district, KwaZulu-Natal, South Africa.
Brief Title: Impact of Immediate Versus South African Recommendations Guided ART Initiation on HIV Incidence
Acronym: TasP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Africa Centre For Health and Population Studies (Other); University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12249 TasP
Record Dates: First submitted 2011-12-20; First posted 2012-01-13 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infection
Keywords: HIV; Prevention; Treatment; South Africa
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate ARV treatment initiation (Experimental): Initiation of ARV treatment regardless of participants's immunological and clinical staging
  Interventions: Drug: Immediate ARV treatment initiation with TDF/FTC/EFV
- South African recommendation guided ARV initiation (Other): HIV-infected individuals will be assessed clinically and immunologically and when eligible for treatment as per South African guidelines will be offered ART
  Interventions: Other: South African recommendation guided ARV (TDF/FTC/EFV) initiation

INTERVENTIONS:
Drug: Immediate ARV treatment initiation with TDF/FTC/EFV — All HIV-infected adults will be offered ART regardless of their immunological and clinical staging.
  The first line regimen proposed will be Atripla (R), a fixed dose combination containing tenofovir disoproxil (245 mg)/emtricitabine (200 mg)/efavirenz (600 mg)(FTC/TDF/EFV). The dosing will be 1 tablet OD.
  Arms: Immediate ARV treatment initiation
Other: South African recommendation guided ARV (TDF/FTC/EFV) initiation — HIV-infected adult participants will be eligible for ART as per the South African guidelines (August 2011) if:
  * CD4 count ≤ 350 cells/mm3 irrespective of clinical symptoms
  * WHO clinical stage 3 or 4 irrespective of CD4 count
  * MDR or XDR TB The first line regimen proposed will be Atripla (R), a fixes dose combination containing tenofovir disoproxil (245 mg)/emtricitabine (200 mg)/efavirenz (600 mg)(TDF/FTC/EFV). The dosing will be 1 tablet OD.
  Arms: South African recommendation guided ARV initiation

SUMMARY:
This trial is evaluating a public health intervention strategy trial which aims to reduce the incidence of HIV at a population-level.

The proposed strategy is a two steps process:

* Extensive HIV counselling and testing, and comprehensive prevention programme among a target population
* Immediate ART initiation after HIV diagnosis, irrespective of CD4 count criteria.

The underlaying trial hypothesis is that HIV testing followed by immediate ART initiation of all HIV-infected individuals will prevent onward transmission and reduce HIV incidence in the population. This is a cluster randomised controlled trial with a total of 22 communities used as the units for randomisation. Enrolment of a population of 22 000 individuals among which 4 400 are expected to be HIV-Infected.

DETAILED DESCRIPTION:
The trial objective is to estimate the effect of ART initiated immediately after HIV diagnosis on the reduction in incidence of new HIV infections in the general population. It will be conducted in two phases:

* First phase: aiming to evaluate the feasibility and acceptability of extensive HIV testing and early ARV treatment initiation on a subset of the target population (Hlabisa sub-district in KwaZulu Natal, South Africa); completion on February 2014.
* Second phase: full implementation of the trial in the target population from May 2014.

The proposed intervention has two components :

* Component 1 "Test": HIV counselling and testing, and comprehensive prevention programme among the entire target population
* Component 2 "Treat": ART treatment initiation for HIV infected individuals following two strategies

  * control group: ART initiation when eligible for treatment as per WHO guidelines
  * intervention group: immediate ART initiation regardless of immunological and clinical staging

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 and more
* Member of a household in the designated cluster within the Hlabisa sub-district of KwaZulu Natal in South Africa
* Able and willing to give written informed consent for trial participation and/or HIV counselling and testing

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28153 (Actual)
Dates: Start 2012-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Uptake of initial and repeat HIV counselling and testing (Feasibility phase) | 14 months
  Percentage of the target population tested for HIV
Uptake of ARV treatment among HIV-infected individuals (Feasibility phase) | 14 months
  Percentage of HIV-infected patients followed-up in the trial clinics receiving ARV treatment when eligible
HIV infection incidence | 4 years after enrolment initiation
  Serology will be done on Dry Blood Spot collected during repeated surveys

SECONDARY OUTCOMES:
Sexual partnerships | Repeated measure every 6 months during follow-up
  Percentage of participants reporting a certain number of sexual partnerships in the last 12 months
Safe sex and condom use | Repeated measure every 6 months during follow-up
  Percentage of participants using a male condom with their partner during the last sexual intercourse
Quality of life | Repeated measure every 6 months during follow-up
  * the EQ-5D scale among the whole sample
  * the Patient Reported Outcomes Quality Of Life specific to HIV (PROQOL-HIV) instrument and the HIV/AIDS stigma instrument for PLWHA (HASI-P) tool among HIV-infected participants
Health care use and health care expenditures | Repeated measure every 6 months during follow-up
  Percentage of participants reporting health care visits (primary care centre, pharmacy, hospitalisation) in the past four weeks and cost incurred
Stigma at community level | Repeated measure every 6 months during follow-up
  Percentage of participants agreeing that people in the community do not blame people for having HIV Percentage of participants agreeing that people in the community avoid people with HIV
Adherence to ART | Repeated measure every 6 months during follow-up
  Measured three-monthly using a visual analogue scale, pill identification test and pill count
Retention | Repeated measure every 6 months during follow-up
  Proportion of HIV-infected participants still under active follow-up in the trial at key timepoints

CONTACTS AND LOCATIONS:
Overall Officials: François Dabis, PhD, Study Chair — INSERM unit 897, ISPED, Université Bordeaux II, France; Marie-Louise Newell, PhD, Study Chair — University of Southamton, United Kingdom; Deenan Pillay, PhD, Study Chair — Africa Centre for Health and Population Studies, University of KwaZullu Natal, South Africa
Locations (1):
- Hlabisa Hospital, Hlabisa, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Iwuji C, Chimukuche RS, Zuma T, Plazy M, Larmarange J, Orne-Gliemann J, Siedner M, Shahmanesh M, Seeley J. Test but not treat: Community members' experiences with barriers and facilitators to universal antiretroviral therapy uptake in rural KwaZulu-Natal, South Africa. PLoS One. 2020 Sep 24;15(9):e0239513. doi: 10.1371/journal.pone.0239513. eCollection 2020. PMID 32970730
- [Derived] Larmarange J, Diallo MH, McGrath N, Iwuji C, Plazy M, Thiebaut R, Tanser F, Barnighausen T, Orne-Gliemann J, Pillay D, Dabis F; ANRS 12249 TasP Study Group. Temporal trends of population viral suppression in the context of Universal Test and Treat: the ANRS 12249 TasP trial in rural South Africa. J Int AIDS Soc. 2019 Oct;22(10):e25402. doi: 10.1002/jia2.25402. PMID 31637821
- [Derived] Perriat D, Plazy M, Gumede D, Boyer S, Pillay D, Dabis F, Seeley J, Orne-Gliemann J; ANRS 12249 TasP Study Group. "If you are here at the clinic, you do not know how many people need help in the community": Perspectives of home-based HIV services from health care workers in rural KwaZulu-Natal, South Africa in the era of universal test-and-treat. PLoS One. 2018 Nov 9;13(11):e0202473. doi: 10.1371/journal.pone.0202473. eCollection 2018. PMID 30412926
- [Derived] Derache A, Iwuji CC, Baisley K, Danaviah S, Marcelin AG, Calvez V, de Oliveira T, Dabis F, Porter K, Pillay D. Impact of Next-generation Sequencing Defined Human Immunodeficiency Virus Pretreatment Drug Resistance on Virological Outcomes in the ANRS 12249 Treatment-as-Prevention Trial. Clin Infect Dis. 2019 Jul 2;69(2):207-214. doi: 10.1093/cid/ciy881. PMID 30321314
- [Derived] Larmarange J, Diallo MH, McGrath N, Iwuji C, Plazy M, Thiebaut R, Tanser F, Barnighausen T, Pillay D, Dabis F, Orne-Gliemann J; ANRS 12249 TasP Study Group. The impact of population dynamics on the population HIV care cascade: results from the ANRS 12249 Treatment as Prevention trial in rural KwaZulu-Natal (South Africa). J Int AIDS Soc. 2018 Jul;21 Suppl 4(Suppl Suppl 4):e25128. doi: 10.1002/jia2.25128. PMID 30027600
- [Derived] Iwuji C, McGrath N, Calmy A, Dabis F, Pillay D, Newell ML, Baisley K, Porter K. Universal test and treat is not associated with sub-optimal antiretroviral therapy adherence in rural South Africa: the ANRS 12249 TasP trial. J Int AIDS Soc. 2018 Jun;21(6):e25112. doi: 10.1002/jia2.25112. PMID 29890048
- [Derived] Iwuji CC, Orne-Gliemann J, Larmarange J, Balestre E, Thiebaut R, Tanser F, Okesola N, Makowa T, Dreyer J, Herbst K, McGrath N, Barnighausen T, Boyer S, De Oliveira T, Rekacewicz C, Bazin B, Newell ML, Pillay D, Dabis F; ANRS 12249 TasP Study Group. Universal test and treat and the HIV epidemic in rural South Africa: a phase 4, open-label, community cluster randomised trial. Lancet HIV. 2018 Mar;5(3):e116-e125. doi: 10.1016/S2352-3018(17)30205-9. Epub 2017 Nov 30. PMID 29199100
- [Derived] Collier D, Iwuji C, Derache A, de Oliveira T, Okesola N, Calmy A, Dabis F, Pillay D, Gupta RK; French National Agency for AIDS and Viral Hepatitis Research (ANRS) 12249 Treatment as Prevention (TasP) Study Group. Virological Outcomes of Second-line Protease Inhibitor-Based Treatment for Human Immunodeficiency Virus Type 1 in a High-Prevalence Rural South African Setting: A Competing-Risks Prospective Cohort Analysis. Clin Infect Dis. 2017 Apr 15;64(8):1006-1016. doi: 10.1093/cid/cix015. PMID 28329393
- [Derived] Iwuji CC, Orne-Gliemann J, Larmarange J, Okesola N, Tanser F, Thiebaut R, Rekacewicz C, Newell ML, Dabis F; ANRS 12249 TasP trial group. Uptake of Home-Based HIV Testing, Linkage to Care, and Community Attitudes about ART in Rural KwaZulu-Natal, South Africa: Descriptive Results from the First Phase of the ANRS 12249 TasP Cluster-Randomised Trial. PLoS Med. 2016 Aug 9;13(8):e1002107. doi: 10.1371/journal.pmed.1002107. eCollection 2016 Aug. PMID 27504637
- [Derived] Orne-Gliemann J, Larmarange J, Boyer S, Iwuji C, McGrath N, Barnighausen T, Zuma T, Dray-Spira R, Spire B, Rochat T, Lert F, Imrie J; ANRS 12249 TasP Group. Addressing social issues in a universal HIV test and treat intervention trial (ANRS 12249 TasP) in South Africa: methods for appraisal. BMC Public Health. 2015 Mar 1;15:209. doi: 10.1186/s12889-015-1344-y. PMID 25880823
- [Derived] Iwuji CC, Orne-Gliemann J, Tanser F, Boyer S, Lessells RJ, Lert F, Imrie J, Barnighausen T, Rekacewicz C, Bazin B, Newell ML, Dabis F; ANRS 12249 TasP Study Group. Evaluation of the impact of immediate versus WHO recommendations-guided antiretroviral therapy initiation on HIV incidence: the ANRS 12249 TasP (Treatment as Prevention) trial in Hlabisa sub-district, KwaZulu-Natal, South Africa: study protocol for a cluster randomised controlled trial. Trials. 2013 Jul 23;14:230. doi: 10.1186/1745-6215-14-230. PMID 23880306